CLINICAL TRIAL: NCT00210288
Title: A Comparative Double Blind Placebo-Controlled Study of Immunogenicity and Safety of Two Doses 10^5 and 10^7 CFU of SC599 Oral Vaccine, a Live Attenuated Shigella Dysenteriae 1 Vaccine Strain in Healthy Human Adult Volunteers
Brief Title: Healthy Adult Volunteer Study for Two Doses of a Shigella Vaccine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institut Pasteur (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: RBM 2004.20
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2018-08-08 (Actual); Status verified 2010-03

CONDITIONS: Shigella Infection
Keywords: Healthy Volunteer; Shigella; Oral Vaccine; Double Blind; Placebo; Immunogenicity; Safety
MeSH Terms: conditions — Dysentery, Bacillary

INTERVENTIONS:
Biological: SC599

SUMMARY:
The purpose of this study is to assess the immune response produced by two doses of SC599 vaccine compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Adult volunteers age 18 to 50
* Signed Informed Consent form following a detailed written explanation of participation in the protocol
* Volunteers who are in good health as determined by medical history, physical examination and clinical judgement
* Volunteers who will be available and "normally reside within the M25" (England) or in Paris and Paris suburb (France) and not leave England or France for the duration of the study
* Women who agree to have a pregnancy test immediately before immunisation and to use effective contraception during the study period
* Volunteers eligible for free NHI treatment (England), volunteers who are covered by social security (France)

Exclusion Criteria:

* Individuals who have hypersensitivity to any component of the vaccines used in this study.
* Individuals who have hypersensitivity to ciprofloxacin
* Individuals who are found to be HIV or HCV antibody positive or Hepatitis B surface antigen positive at the time of initial screening
* Individuals who are found to have HLA-B27 tissue type at the time of initial screening
* Individuals with a known or suspected history of gastrointestinal disease or abnormality
* Concomitant therapy with antibiotics, iron, zinc, H2-receptor antagonists or proton pump inhibitors
* Individuals who have received any vaccine against Shigella or had proven or suspected shigellosis (bloody diarrhoea with fever) within 6 months prior to study entry
* Individuals with a significant level of immunity against Shigella detected at the screening visit (defined as serum ELISA anti-LPS IgG antibody titre greater than 3 S.D. above the mean background activity of a bank of healthy human sera)
* A Clinically significant amount of protein or haemoglobin in the urine sample at the screening visit
* A Clinically significant abnormality in the haematological or biochemical assays (an abnormal value will be defined by the ranges quoted in each centre) at the screening visit
* A positive Shigella stool culture at the screening visit
* Individuals with a known impairment of immune function or those receiving immunosuppressive therapy (including systemic corticosteroids). Inhaled or topical steroid preparation are not a non-inclusion criterion
* Individuals with acute infections (including fever > 37.5°C oral temperature)at the time of immunisation or any chronic disease
* Women capable of becoming pregnant who do not agree to have pregnancy testing before immunisation, or who do not agree to take effective contraception during the study period
* Breastfeeding women
* Individuals with a current problem with substance abuse or with a history of substance abuse which in the opinion of the investigator, might interfere with participation in the study
* Individuals with any condition which, in the opinion of the investigator, might interfere with the evaluation with the study objectives
* Individuals who have received an investigational product within 30 days prior to entry
* Individuals who cannot read, speak fluent French or English according to the investigational site setting
* Individuals who are planning to leave England or France prior to the end of the study period or who are likely not to complete the study
* Individuals who have persons living with them who in the opinion of the investigator may be at risk of disease if exposed to the vaccine strain or whose occupation may bring them into contact with persons at risk of disease or who are food handlers by occupation
* Individuals with close household contact with child younger than 5 years or a person with immunodeficiency

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 111 (Estimated)
Dates: Start 2005-05; Primary Completion 2006-09 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Immune response assessed by the proportion of Immunoglobulin A (IgA) anti-Lipopolysaccharide (LPS) Antibody-Secreting Cells (ASC) responders.

SECONDARY OUTCOMES:
1) Immune Response:
-Proportion of volunteers who have a B subunit antibody response
-Proportion of volunteers who have a LPS response
2) SC599 Shedding
-Proportion of volunteers who will excrete the vaccine strain and by the duration of the SC5999 shedding, defined as the time (days) between the first an last stool that were positive for SC599.
3) Safety Assessment
-The safety will be evaluated by the proportions of clinical and biological adverse events. Illness after vaccination will be defined as either diarrhoea or fever.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Odile Launay, MD, Principal Investigator — Hôpital Cochin - Bâtiment Modulaire, France; Dr David Lewis, MD, Principal Investigator — St George's Hospital Vaccine Institute, UK
Locations (2):
- CIC de Vaccinologie Cochin Pasteur, Paris, France
- Dept of Cellular and Molecular Medicine, St George's Hospital Vaccine Institute, London, United Kingdom